CLINICAL TRIAL: NCT06411145
Title: A Prospective, Multicenter Trial to Evaluate Efficacy and Safety of Cenegermin-bkbj (20 mcg/mL) Ophthalmic Solution on Corneal Thickness Via Anterior Segment Optical Coherence Tomography (AS-OCT) in Stage 3 Neurotrophic Keratitis
Brief Title: Open-label Trial to Evaluate Efficacy and Safety of rhNGF on Corneal Thickness Via AS-OCT in Neurotrophic Keratitis
Acronym: IMAGO
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was withdrawn prior to enrolling subjects due to realignment of strategic priorities.
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGF0223
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Neurotrophic Keratitis; Neurotrophic Keratopathy; Corneal Ulcer
Keywords: stage 3 keratitis; cenegermin-bkbj; OXERVATE®; rhNGF
MeSH Terms: conditions — Corneal Ulcer; Keratitis | interventions — cenegermin

STUDY DESIGN:
Intervention Model Description: Cenegermin-bkbj (20 mcg/mL) ophthalmic solution contained in a multiple-dose vial. The topical drops are administered 6 times/day for a 6-week course.
Masking Description: This is an open label study, hence masking is not applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cenegermin-bkbj (Experimental): cenegermin-bkbj (20 mcg/mL) ophthalmic solution on corneal thickness administered as topical drops via anterior segment optical coherence tomography (AS-OCT), where cenergermin-bkbj stands for Topical Recombinant Human Nerve Growth Factor (rhNGF). Cenegermin-bkbj, the active ingredient of OXERVATE® 0.002% (20 mcg/mL) cenegermin-bkbj ophthalmic solution, is structurally identical to the human nerve growth factor (NGF) protein made in ocular tissues.
  Interventions: Drug: OXERVATE® 0.002%

INTERVENTIONS:
Drug: OXERVATE® 0.002% — Cenegermin-bkbj (20 mcg/mL) is an ophthalmic solution contained in a multiple-dose vial. The topical drops are administered 6 times/day for a 8-week course.
  Other Names: cenegermin-bkbj

SUMMARY:
Primary Objective:

To assess the efficacy of cenegermin-bkbj (20 mcg/mL) ophthalmic solution on overall corneal thickness via AS-OCT in patients with stage 3 neurotrophic keratitis with respect to change from baseline at weeks 4, 8, and 16.

Secondary Objectives:

To assess the effects of cenegermin-bkbj (20 mcg/mL) ophthalmic solution on corneal stromal thickness via AS-OCT in patients with stage 3 neurotrophic keratitis with respect to change from baseline at weeks 4, 8, and 16.

To assess the effects of cenegermin-bkbj (20 mcg/mL) ophthalmic solution on corneal stromal reflectivity via AS-OCT in patients with stage 3 neurotrophic keratitis with respect to change from baseline at weeks 4, 8, and 16.

To assess the effects of cenegermin-bkbj (20 mcg/mL) ophthalmic solution on corneal sensitivity via Cochet-Bonnet aesthesiometer in the center of the lesion with respect to change from baseline at weeks 4, 8, and 16.

DETAILED DESCRIPTION:
This clinical study is a prospective, open-label, interventional, multicenter study of 8 weeks of treatment with 8 weeks of follow-up after treatment to evaluate the efficacy of cenegermin-bkbj (20 mcg/mL) ophthalmic solution on corneal thickness and stromal clarity via AS-OCT in patients with stage 3 neurotrophic keratitis.

The study will be a total of 16 weeks in duration: an optional screening period of up to 2 weeks, followed by an 8-week treatment period and an 8-week follow-up period. At Visit 1.2 (Baseline and Study Product Dispense, Day -1), patients meeting the entry criteria for this study will be assigned to treatment with cenegermin-bkbj (20 mcg/mL) ophthalmic solution (which will be known as Study Product) beginning the morning following that visit, or Day 0.

After completion of the Treatment Period, all patients who do not meet deterioration or no improvement criteria will continue to be followed for an additional 8-week Follow-Up Period.

At any time during the study, patients may be seen for additional unscheduled visits as deemed necessary by the Investigator.

For patients who are prematurely discontinued from the study at any point, an exit examination should be completed which represents the next data collection visit in the study timeline. Once exited, the Investigator should direct patients for further treatment as appropriate. Patients in this study who are prematurely discontinued before completion of 8 weeks of treatment with cenegermin-bkbj (20 mcg/mL) ophthalmic solution will continue to be followed throughout the remainder of the study period, if able.

To minimize risk of bias, all images will be assessed at an independent central reading center (CRC). The study site will acquire the images and perform a quality check; however, no analysis is required to be conducted by the Investigator on site.

Visits list:

1. Visit 1.1- Screening Visit (Day -14 to -1)
2. Visit 1.2- Baseline Visit and Study Product Dispensation (Day -1)
3. Treatment Period (Weeks 1-8)
4. Visit 2- Study Product Dispensation (Day 14 ± 3 days)
5. Visit 3- Mid-Treatment Week 4 Evaluation and Study Product Dispensation(Day 28 ± 3 days)
6. Visit 4- Study Product Dispensation Visit (Day 42 ± 3 days)
7. Visit 5- End-of-Treatment Week 8 Evaluation (Day 56 ± 3 days)
8. Follow-Up Period (Weeks 9-16)
9. Visit 6- Final Follow-Up Week 16 Evaluation (Day 112 ± 3 days)

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥18 years of age at time of screening.
2. Patient must be stage 3 NK in the study eye defined by the Mackie Criteria at baseline (Appendix 4).
3. Evidence of decreased corneal sensitivity in the study eye as measured by Cochet-Bonnet esthesiometry (≤4 cm in the center of the neurotrophic lesion) at baseline.
4. Patients who have only one functional eye can be included if they meet all the criteria above and per the Investigator's discretion are proper candidates to designate the one functional eye as the study eye.
5. Self-retaining amniotic membrane or any other amniotic topical product may be used prior to baseline visit (Visit 2) but should be removed or fully dissolved by the baseline measurements.
6. Patients must have the ability and willingness to comply with study procedures and study product dosing as described in the protocol.
7. Only patients who satisfy all informed consent requirements may be included in the study. The patient and/or his/her legal representative must read, sign, and date the Institutional Review Board (IRB)-approved informed consent document before any study-related procedures are performed.

Exclusion Criteria:

1. In the opinion of the Investigator, evidence or confirmed culture of an active ocular infection (bacterial, fungal, protozoal) in either eye at the time of screening or baseline.
2. Evidence of a necrotizing herpetic ulcer in either eye at the time of screening or baseline.
3. Active or severe corneal/ocular inflammation that requires continuous medical therapy throughout the duration of the treatment, including eyelid-based disorders such as severe MGD or blepharitis.
4. Patients with posterior one-third corneal involvement or if posterior one-third of cornea becomes involved during the time between screening and baseline measurements, or at the Investigator's discretion is close to perforation.
5. Patients who have excessive, pre-existing corneal opacification.
6. Any of the following within 90 days of study enrollment:

   1. Treatment with Botox (botulinum toxin) injections in the study eye to induce pharmacologic blepharoptosis
   2. Treatment with intravenous chemotherapy for oncologic pathology
7. Patients who have punctal occlusion planned within the study period. Patients who have undergone punctal occlusion prior to entry into the study are eligible for enrollment provided that the punctal occlusion is maintained during the study period. If a punctal plug falls out of the study eye during the study, it must be reinserted within 7 days of discovery via examination by the Investigator.
8. Anticipated need to use therapeutic contact lenses, contact lens wear for refractive correction, or scleral contact lenses during the treatment period in the study eye.
9. Patients with eyelid or neuromuscular abnormality that may alter eyelid function or closure, thereby increasing exposure; this includes but is not limited to blepharospasm, cranial nerve palsy or paresis, entropion, ectropion, or floppy eyelid syndrome.
10. Previously been treated with OXERVATE®
11. Ocular surgeries (including but not limited to LASIK, PRK, tube shunt/trabeculectomy, cataract surgery) within the last 6 months.
12. History of corneal stromal surgery, including anterior lamellar keratoplasty (ALK), deep anterior lamellar keratoplasty (DALK), and penetrating keratoplasty (PKP) within 12 months of screening visit
13. Female patients who are pregnant or lactating at study screening or baseline, or those who are planning pregnancy during the period of study.
14. Premenopausal females not using a medically acceptable form of birth control (abstinence, pharmaceutical contraception, intrauterine device, surgically sterilized) during the treatment period.
15. History of drug addiction or alcohol abuse documented within the past 2 years.
16. Patients who are active smokers shall be excluded.
17. Actively participating in a clinical trial at time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-26 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Change in overall corneal thickness via AS-OCT from baseline to weeks 4, 8, and 16. | weeks 4, 8, and 16.
  The changes from baseline in corneal thickness via AS-OCT from baseline to weeks 4, 8, and 16 will be analyzed by means of an adjusted longitudinal regression model

SECONDARY OUTCOMES:
Change in corneal stromal thickness via AS-OCT from baseline to weeks 4, 8, and 16. | weeks 4, 8, and 16
  the effects of cenegermin-bkbj (20 mcg/mL) ophthalmic solution on corneal stromal thickness via AS-OCT will be assessed in patients with stage 3 neurotrophic keratitis
Change in stromal reflectivity via AS-OCT from baseline to weeks 4, 8, and 16 | weeks 4, 8, and 16
  corneal stromal reflectivity via AS-OCT in patients with stage 3 neurotrophic keratitis will be assessed
Change in corneal sensitivity within lesion area via Cochet-Bonnet from baseline to weeks 4, 8, and 16. | weeks 4, 8, and 16
  Change in corneal sensitivity within lesion area via Cochet-Bonnet aesthesiometer will be assessed
Frequency and severity of TEAE throughout the study until the FU week 16 assessment (Day 112 +/- 3) | Throughout the study until Day 112 +/- 3
  AEs will be coded by preferred term and system organ class by using the latest version of the Medical Dictionary for Regulatory Activities AEs will be summarized overall, by severity, and by relationship to study product. Serious AEs and AEs leading to discontinuation of study product will also be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Kligman, MD, Principal Investigator — SightMD, New York, New York

IPD SHARING:
Plan to Share IPD: No